CLINICAL TRIAL: NCT03756519
Title: Determining the Effects of Adding Exercise to Usual Care for Recent Onset Low Back Pain in the Emergency Department: A Randomized Controlled Trial
Brief Title: The Effect of Exercise on Recent Onset Low Back Pain in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Jordan Miller, PT, PhD, Assistant Professor, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REH-715-18
Record Dates: First submitted 2018-04-19; First posted 2018-11-28 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Low Back Pain
Keywords: acute; exercise; emergency department
MeSH Terms: conditions — Low Back Pain; Motor Activity; Emergencies | interventions — Exercise; Hot Temperature

STUDY DESIGN:
Intervention Model Description: The patient will be partially blinded by our not providing full details on the two interventions being studied. Participants will be instructed that, "Participants in this study will be randomized (chosen as by a coin flip) to receive one of two different types of advice and instruction on maintaining mobility and performing exercise."
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Participants in the exercise intervention arm will receive the usual care protocol plus a standardized, evidence informed exercise intervention provided by trained physiotherapy students. The exercise intervention will begin with a brief assessment to rule out contraindications to exercise and to identify any directional preferences (e.g. pain with lumbar flexion and relief with extension). The PT will then be taught four standardized exercises: the pelvic tilt exercise, a rotational exercise, a tailored graded walking program taking into account the current abilities of the patient, and an exercise based on the directional preference of the individual. These will be re-enforced with a handout including the rationale, instructions and dosage recommendations for the exercises.
  Interventions: Behavioral: Exercise; Behavioral: Advice to stay active and engaged in usual activities.; Behavioral: Advice on use of ice or heat; Other: Advise regarding use of medications
- Usual care (Active Comparator): Our usual care protocol was developed based on 30 responses to an 18 item survey of Queen's Department of Emergency Medicine physicians. Three themes emerged as interventions most commonly used. Each of these strategies has evidence for small, but positive treatment effects and low risk of harms: 1) advice to stay active and engaged in usual activities, 2) use of ice or heat to manage pain, and 3) recommendation for analgesia using NSAIDs if needed and appropriate.
  Interventions: Behavioral: Advice to stay active and engaged in usual activities.; Behavioral: Advice on use of ice or heat; Other: Advise regarding use of medications

INTERVENTIONS:
Behavioral: Exercise — A standardized exercise program tailored to the individual based on their directional preferences and current functional abilities.
  Arms: Exercise
Behavioral: Advice to stay active and engaged in usual activities. — Participants will be advised that staying physically active and continuing to participate in usual activities improves recovery. This verbal advice will be reinforced with a written handout.
Behavioral: Advice on use of ice or heat — Participants will be advised on the appropriate use of ice or heat to manage pain. This verbal advice will be reinforced with a written handout.
Other: Advise regarding use of medications — Participants will receive education regarding the use of non-steroidal anti-inflammatory medications (NSAIDs) for pain relief, if needed and if the patient is appropriate for NSAIDs. Information regarding specific recommended doses, potential benefit and risk will be discussed.

SUMMARY:
Low back pain (LBP) is the leading contributor to years lived with disability and an important contributor to healthcare costs and time off work. Exercise is effective for chronic low back pain, but there is a lack of evidence to inform whether exercise in the emergency department is effective for people with acute low back pain. This randomized controlled trial will evaluate the effectiveness of a brief exercise intervention provided in the emergency department for people with recent onset low back pain. People with acute low back pain (<1 week) will be randomly assigned to either usual care or to usual care plus a brief exercise intervention delivered by trained physiotherapy students. The study will evaluate the impact of the added exercises on self-reported disability (primary outcome), pain intensity, global rating of change, patient satisfaction, and adverse events. In addition, we will pilot data collection related to return to work, healthcare utilization, and cost effectiveness outcomes to determine the feasibility of conducting a future trial with additional patient participants required to evaluate these outcomes. Outcomes will be evaluated at baseline, 48-72 hours, 1-week, 1-month, and 3-months from their initial emergency department visit. The results of this study have the potential to inform emergency department management of acute low back pain.

DETAILED DESCRIPTION:
Low back pain (LBP) is the leading contributor to years lived with disability and an important contributor to healthcare costs and time off work. Exercise is effective for chronic low back pain, but there is a lack of evidence to inform whether exercise in the emergency department is effective for people with acute (<1 week) low back pain.

The objectives of this randomized controlled trial are:

1. To determine the effectiveness of an exercise intervention delivered in the ED in comparison to usual ED care on pain, function, global rating of change, patient satisfaction, and adverse effects in adults with recent onset LBP (< 1 week).
2. To determine the feasibility of a future RCT to evaluate the effects of the ED exercise intervention on return to work outcomes, health care utilization, and cost-effectiveness in comparison to usual care.

The investigators hypothesize that an exercise intervention in the ED will improve pain, function, global rating of change, and patient satisfaction in comparison to usual ED care with no difference in adverse effects.

Design: A randomized controlled trial (RCT) with two parallel arms (exercise and usual care).

Blinding: The patient will be partially blinded by our not providing full details on the two exercise approaches being studied. The health care providers delivering the interventions will not be blinded due to the nature of the intervention. However, research assistants administering the outcome measures will be blinded. The outcomes assessed are objective measures assessed using an online survey tool that will be free of assessor bias.

Randomization and allocation concealment: Participants will be randomized in a 1:1 ratio to exercise or usual care groups by an independent statistician using a computerized random number generator. The random allocation will be placed in sequentially numbered opaque envelopes. The envelopes will be opened by the RA after completion of baseline assessment.

Patient enrollment: Consecutive patients with acute LBP who are seeking urgent care at Kingston General Hospital Emergency Department (ED) and Hotel Dieu Hospital Urgent Care Clinic (UCC) will be invited to participate over a 4-month period May 1 through August 31, 2018). ED based research staff will screen patients for willingness to be invited to participate when they arrive at the ED. These staff will then invite participation once the physician assessment is complete and eligibility criteria are reviewed.

Inclusion criteria: English speaking adults (18-65 years) with recent onset LBP (<1 week).

Exclusion criteria: people with subacute/chronic LBP, previous episode of back pain in the past 3 months, fracture, previous back surgery, red flags (e.g. urinary retention, bilateral or multilevel neurological impairment), traumatic mechanism of injury (fall >3m or 3 steps, MVC >100km/h).

Assessment and outcome measures: All measures will be collected using Qualtrics, a secure online database, at baseline, 48-72 hours, 1-week, 1-month, and 3-months.

Baseline factors used to describe the population: age, gender, duration of back pain (hours), whether there have been previous episodes of back pain, whether or not the participant has pain in other areas of the body, medications, comorbidities, work status prior to onset of back pain, and current work status.

Objective #1: Individual health outcomes will be collected using validated tools described under the outcomes assessed.

Objective #2: This study design will not have adequate power or long-term follow-ups required to adequately evaluate return to work, healthcare use, and cost-effectiveness. The investigators plan to pilot the use of these outcomes to determine the feasibility of conducting a future trial to evaluate these outcomes.

Analysis: For objective #1, Repeated-measure linear mixed models will be used to assess the effect of treatment (exercise versus usual care) on our primary (disability) and secondary (pain, global rating of change, patient satisfaction, adverse effects) outcomes at all time-points (48-72 hours, 1-week, 1- and 3-months). A difference of 2 on the NPRS36 and 3 points on the RMDQ37 will be considered clinically meaningful. For objective #2, all feasibility outcomes will be reported descriptively and analyzed qualitatively as recommended by methods and reporting guidelines for pilot and feasibility studies.

Sample size: The investigators searched one year of ED and UCC records to identify LBP patients eligible for this study. 2000 patients/year attended for back pain with > 500 during our four-month recruitment period. Of these, a chart review suggests 43% of these met our eligibility criteria. Based on past trials in these settings, we expect at least 50% will consent resulting in a sample size of 107+. This will achieve over 90% power to detect a minimally important difference of 3 points on the RMQ, using a two-sided α=0.05 and assuming a standard deviation of 6.2 points and accounting for a 10% loss to follow-up. This will also provide an adequate sample to assess the secondary feasibility objectives.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Adults (18-65 years)
* Recent onset low back pain (<1 week)

Exclusion Criteria:

* Subacute/chronic LBP (> 1week)
* Previous episode of low back pain in past 3 months
* fracture
* previous back surgery
* urinary retention
* saddle anaesthesia
* bilateral or multilevel neurological impairment
* traumatic mechanism of injury (fall >3m or 3 steps, MVC >100km/h).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Self-reported disability | Change from baseline to 3-months with repeated measures at baseline, 1-week, 1-month, 3-months and a primary comparison at 1-week
  Roland Morris Questionnaire (0-24, higher represents greater disability)

SECONDARY OUTCOMES:
Pain Intensity currently | Change from baseline to 3-months with repeated measures at baseline, 1-week, 1-month, 3-months and a primary comparison at 1-week
  Numeric pain rating scale (0-10, higher represents greater pain intensity)
Pain intensity on average over past 24-hours | Change from baseline to 3-months with repeated measures at baseline, 1-week, 1-month, 3-months and a primary comparison at 1-week
  Numeric pain rating scale (0-10, higher represents greater pain intensity)
Pain intensity at its worst over the past 24-hours | Change from baseline to 3-months with repeated measures at baseline, 1-week, 1-month, 3-months and a primary comparison at 1-week
  Numeric pain rating scale (0-10, higher represents greater pain intensity)
Pain intensity at its least over the past 24-hours | Change from baseline to 3-months with repeated measures at baseline, 1-week, 1-month, 3-months and a primary comparison at 1-week
  Numeric pain rating scale (0-10, higher represents greater pain intensity)
Global rating of change | 1-week, 1-month, 3-months with a primary comparison at 1-week
  Perceived change in function (-5 to +5, higher represents greater improvement in function)
Patient satisfaction | 1-week, 1-month, 3-months with a primary comparison at 1-week
  Satisfaction with healthcare received (-5 to +5, higher represents greater satisfaction with care)
Adverse effects | 1-week, 1-month, 3-months with a primary comparison at 1-week
  Self-reported adverse effects of treatment
Treatment fidelity | At initial visit
  A fidelity checklist performed by the physiotherapy students carrying out the intervention will be included as a process outcome.
Recruitment rate (to determine feasibility for future trial on healthcare utilization, cost-effectiveness and return to work) | Recruitment rate over 4 month period
  Rate of recruitment (number of participants/week over recruitment period)
Retention rate (to determine feasibility for future trial) | Baseline, 1-week, 1-month, 3-months with a primary time-point of 3-month follow-up
  Rate of assessment completion
Work status - working or not working (piloted to determine the feasibility of conducting a future trial evaluating return to work outcomes) | Baseline, 1-week, 1-month, 3-months with a primary time-point of 1-week
  Work status (working/not working)
Work status - full or part time (piloted to determine the feasibility of conducting a future trial evaluating return to work outcomes) | Baseline, 1-week, 1-month, 3-months with a primary time-point of 1-week
  Work status (full/part-time)
Work status - full or modified duties/hours(piloted to determine the feasibility of conducting a future trial evaluating return to work outcomes) | Baseline, 1-week, 1-month, 3-months with a primary time-point of 1-week
  Work status - full/modified duties or hours
Work status - hours worked (piloted to determine the feasibility of conducting a future trial evaluating return to work outcomes) | Baseline, 1-week, 1-month, 3-months with a primary time-point of 1-week
  Number of hours worked in past seven days.
Healthcare utilization (piloted to determine the feasibility of conducting a future trial evaluating healthcare utilization) | 1-week, 1-month, 3-months with a primary time-point of 3-months
  Self-report questoinnaire asking patient to report primary care visits, emergency room visits, hospitalizations, surgeries, consultations with other health care providers (e.g. physiotherapists, chiropractors, physician specialists, diagnostic imaging (e.g. x-ray, CT scan, MRI), and medication
Costs (piloted to determine the feasibility of conducting a cost-effectiveness analysis in a future trial) | All costs incurred between baseline and 3-month follow-up will be calculated
  Includes all healthcare costs as well as societal costs using a human capital approach
Quality of life (piloted to determine feasibility of performing cost-effectiveness analysis in a future trial) | Change from baseline to 3-months with repeated measures at baseline, 1-week, 1-month, 3-months and a primary time-point of 3-months
  EuroQOL 5D-5L (0-100 with greater score indicating greater quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Miller, PhD, Principal Investigator — Queen's University; Robert Brison, MD, Principal Investigator — Kingston Health Sciences Center and Queen's University; Elizabeth Blackmore, MD, Principal Investigator — Kingston Health Sciences Center
Locations (1):
- Kingston Health Sciences Center - Kingston General Hospital and Hotel Dieu Hospital Sites, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No